CLINICAL TRIAL: NCT03264677
Title: An 8-week Full Face HUT Design, Single Center, Double Blinded, Controlled and Randomized Study to Evaluate Different Product Regimens' Performance on Protecting Skin With Resilience Under Tracked City Environmental Aggressors
Brief Title: An 8-week Full Face HUT Clinical Trial for HydroBoost (2.0/3.0)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Pte Ltd (Industry)
Collaborators: Shanghai Skin Disease Hospital (Unknown); Shanghai China-Norm Management Consulting co.,LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CO-170223145432-SACT
Record Dates: First submitted 2017-07-24; First posted 2017-08-29 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Adult Skin Healthy Signs
Keywords: 8-week HUT; Hydro Boost; Skin healthy signs; Environmental aggressors; Cosmetic

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly and evenly divided into 3 groups (approx. 40 subjects per group) with different facial care regimens during the 8-week home use study.
  Group 1: NTG Hydro Boost Gelee Milk Cleanser + NTG Hydro Boost Kiwi Water Gel Group 2: NTG Hydro Boost Gelee Milk Cleanser + NTG Hydro Boost Water Gel Group 3: NTG Hydro Boost Gelee Milk Cleanser + NTG Hydro Boost Extra Dry Emulsion
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Since this will be a blind study, the product randomization codes will be generated by study team member different from Study Manager, Study Director, Principle Investigator and any data producers or influencer. The product randomization codes and the corresponding product information (i.e. product name, formula number, batch number, manufacturing/expiry date, etc.) will be sealed in an envelope and before study filed work complete kept by PI until there is a unblinding needs due to medical emergency or report drafting.
  In this study, in total 4 IPs include 3 facial creams and 1 facial cleanser will be evaluated. Subjects will be assigned to 3 groups randomly and evenly with different facial product regimens (one cleanser + one cream). The product regimens will be applied on the whole face for on-site study and the 8-week HUT. For each subject, left or right cheek area will be randomly chosen as experimental area for evaluation and middle upper chest will be the untreated control area
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): NTG Hydro Boost Gelee Milk Cleanser + NTG Hydro Boost Kiwi Water Gel
  Interventions: Combination Product: Group 1
- Group 2 (Experimental): NTG Hydro Boost Gelee Milk Cleanser + NTG Hydro Boost Water Gel
  Interventions: Combination Product: Group 2
- Group 3 (Experimental): NTG Hydro Boost Gelee Milk Cleanser + NTG Hydro Boost Extra Dry Emulsion
  Interventions: Combination Product: Group 3

INTERVENTIONS:
Combination Product: Group 1 — NTG Hydro Boost Gelee Milk Cleanser + NTG Hydro Boost Kiwi Water Gel
  Other Names: HB Cleanser+Kiwi Water Gel
  Arms: Group 1
Combination Product: Group 2 — NTG Hydro Boost Gelee Milk Cleanser + NTG Hydro Boost Water Gel
  Other Names: HB Cleanser+HB Water Gel
  Arms: Group 2
Combination Product: Group 3 — NTG Hydro Boost Gelee Milk Cleanser + NTG Hydro Boost Extra Dry Emulsion
  Other Names: HB Cleanser+HB ED Emulsion
  Arms: Group 3

SUMMARY:
* To investigate the product regiments' performance on moisturization related skin healthy signs (skin moisturization, barrier function, elasticity, translucency, roughness and skin conditions) through instrumental evaluation, clinical grading and self-assessment before, during and after 8 weeks' home usage under city environmental aggressors (Sun, change of temperature and humidity, wind and air pollution) among 3 product regimens and Non-treatment control;
* To explore the linkage among products efficacy, ambient aggressors, and life habits;
* To investigate product regimens' tolerance and safety via Home Use Test;
* To collect skin microflora/microbiome samples for potential research on skin microbiome distribution change as impacted by product application and/or environmental aggressors change (data will be analyzed and reported separately).

DETAILED DESCRIPTION:
This is a single center, double blinded, controlled and randomized 8-week home use clinical trial.

Subjects will be randomly and evenly divided into 3 groups (40subjects/group) with different facial care regimens during the 8-week home use study.

Group 1: NTG Hydro Boost Gelee Milk Cleanser + NTG Hydro Boost Kiwi Water Gel Group 2: NTG Hydro Boost Gelee Milk Cleanser + NTG Hydro Boost Water Gel Group 3: NTG Hydro Boost Gelee Milk Cleanser + NTG Hydro Boost Extra Dry Emulsion There will be a 3-day wash-in period after subject's enrollment. During the period, no product will be allowed to be applied on the face and upper chest but only water washes twice per day in the morning and evening for 3 days before baseline (BL) measurement.

After baseline (BL) measurement, the product regimens will be applied on face at site under site instruction according to the randomization. Measurements will be taken at 2-4 hours and 8 hours after product regimens' application. Upper chest area will be measured as no treatment control.

A set of product regimen includes a facial cleanser and a facial cream will be distributed to each subject according to grouping and applied on the face at home for 8 weeks. Both cleanser and cream products will be applied twice a day in the morning and evening on the whole face. For the upper chest area, use water wash only twice per day in the morning and evening, no any other product is allowed.

The usage of assigned product regimens will be discontinued after 8-week home use, no any other product is allowed but only water wash twice per day in the morning and evening on both face and upper chest for 3 days (regression period).

Subjects will not be allowed to use sunscreen, makeup and any other cosmetic products on face and upper chest during the study period.

Subjects will visit the site at Screening (-3D), Baseline (BL), 1-week (1W), 4-week (4W), 8-week (8W) and 8-week+3-days (+3D) for measurements.

ELIGIBILITY:
Inclusion Criteria

1. Chinese Females aged 18 - 40 years old in good physical and mental condition;
2. Self-perceived dry facial skin without lesions. Corneometer score ≤35 arbitrary units on both sides of cheek areas;
3. Having daily routine skin exposure (out-door activities) to city environmental challenge and having concern on its impact to healthy skin signs (e.g. Smoothness, Firmness, Translucency, Trouble (pimple, acne) free, Plumpness, etc.);
4. Willing to stay in Shanghai City during the whole study period without travel plan;
5. Having mild to moderate pre-aging sign, e.g. fine line, roughness when skin is dry. Having skin dullness concern on the face;
6. Non-regular body moisturizer user. Expose the upper-chest site during study;
7. Willing to comply with the study instruction (see Appendix IX);
8. Agree to use only water to wash face and upper chest, avoid using any cosmetic products (include but not limited to: wash/ soap/ moisturizer/ toner/ sparge/ sunscreen/ oil/ (water) mask/ scrub/ makeup/ fragrance/ light treatment/ massage, etc.) in the evening before each visit day. No washing on face and upper chest and no product application at home in the morning of the visit day. Subjects will wash the test areas when arrive the test site according to the site instruction;
9. After enrollment, there will be a 3-day wash-in period, during which subjects agree to use water only to wash the face and upper chest twice per day in the morning and evening. Avoid using any cosmetic products as listed in above item 8 in both test areas;
10. Then an 8-week home use period will follow, during which subjects agree to use the assigned product regimens (facial cleanser and facial cream) on face twice per day in the morning and evening. Use water only to wash the upper chest twice per day in the morning and evening. Avoid using any cosmetic products as listed in above item 8 in both test areas;
11. After the 8-week home use of the assigned product regimens, subjects will stop using the products for 3 days (Regression period). Subjects agree to use water only to wash the face and upper chest twice per day in the morning and evening during the period. Avoid using any cosmetic products as listed in above item 8 in both test areas;
12. Generally in good health based on medical history reported by the subject;
13. Female subjects must meet one of the following criteria:

    * Is not of child-bearing potential or is in a monogamous relationship with a partner who is not of child-bearing potential, meaning the subject and/or partner:

      * Is post-menopausal (amenorrhea for at least 1 year),
      * Had a surgical sterilization (e.g., vasectomy that has been confirmed effective by sperm count check, tubal occlusion, hysterectomy, bilateral oophorectomy or salpingectomy)
    * Must agree to practice a medically acceptable form of birth control during the study and for 30 days after study completion. Female subjects must have used such birth control for at least 3 months prior to study start. Medically acceptable forms of birth control that may be used by the subject and/or partner include:

      * Established use of hormonal methods of contraception (oral, injected, implanted, hormone patch or vaginal ring).
      * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps),
      * Intrauterine device or intrauterine system,
      * Abstinence from intercourse that could cause pregnancy. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
14. Is not a ward of the court or deprived from liberty by a judiciary or administrative decision;
15. Able to read, write, speak and understand Chinese language or able to speak and understand Chinese language and accompanied by an impartial witness who can read, write, speak and understand Chinese language;
16. Individual that has signed the Consent for Photograph Release (7-8 subjects/group) and ICD including portable tracker using and reporting as instruction;

Exclusion Criteria

1. Participated in any cosmetic clinical test involving facial and/or body product application within 3 months before enrollment.
2. Has known allergies or adverse reactions to common topical skincare products;
3. Presents with a skin condition that may influence the outcome of the study (e.g., psoriasis, eczema, melanomas), primary/secondary lesions on test sites (e.g. erythema, scars, ulcers, vesicles);
4. Has a self-reported uncontrolled metabolic condition or disease, such as diabetes, hypertension, hyper/hypothyroidism, hypercholesterolemia, asthma, epilepsy, etc. Individuals with a controlled health condition may also be excluded from the study at the discretion of the PI, if medically qualified, or the designated study physician;
5. Is taking medication for a chronic condition (e.g., insulin, antihistamines, steroidal and non-steroidal anti-inflammatory drugs, antibiotics, etc.) or is taking any other medication that could influence the study results and/or affect the individual's safety, within 30 days before inclusion or during the study;
6. Is taking immunosuppressive drugs within 3 months before inclusion and during the study;
7. Has a history of or concurrent health condition/situation which, in the opinion of the PI, if medically qualified, or the designated study physician, may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study;
8. Is simultaneously participating in any other type of clinical study;
9. Is an employee/contractor or immediate family member of the PI, Study Site staff or Sponsor.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Chinese Females
Enrollment: 122 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Skin surface moisture content | 9 weeks
  Skin surface moisture content is measured by skin capacitance measurement.

SECONDARY OUTCOMES:
Quality of Life | 9 weeks
  In this study, an evaluation tool will be used to measure and quantify skin dryness related Quality of Life (QoL) attributes, to get an understanding of the improvement (related to moisturization benefits) after treatment of skin care regimens
Subject Self-assessment | 9 weeks
  Subject self-assessment Questionnaire (QN) on product performance
Temperature | 9 weeks
  Individual temperature measured by portable environmental tracker
Humidity | 9 weeks
  Individual humidity measured by portable environmental tracker
PM 2.5 | 9 weeks
  Individual PM 2.5 measured by portable environmental tracker
Skin microbiome | 9 weeks
  To collect skin microflora/microbiome samples for potential research on skin microbiome distribution change as impacted by product application and/or environmental aggressors change.
Life habits | 9 weeks
  Subject's life pattern captured by diary.
Skin barrier function | 9 weeks
  TEWL
Skin elasticity | 9 weeks
  The mechanical property of the epidermis is measured by a non-invasive, in vivo suction skin elasticity meter.
Skin roughness | 9 weeks
  Skin roughness measurement via skin surface imaging
Skin translucency | 9 weeks
  Many common materials transmit and scatter light but are neither transparent or opaque. Such materials are described as translucent and the degree of translucency depends on the absorption and scattering coefficients of the material. In this study, the degree of skin translucency is quantified by the rate of lateral scatter of light and the total amount of backscattered light, which captured by a non-invasive Translucency Meter probe.
Skin deep layer moisture content | 9 weeks
  Skin deep layer moisture content by measuring skin dielectric constant.
Skin firmness | 9 weeks
  Dermatologist grading of skin firmness
Skin elasticity | 9 weeks
  Dermatologist grading of skin elasticity
Skin radiance | 9 weeks
  Dermatologist grading of skin radiance
Skin smoothness | 9 weeks
  Dermatologist grading of skin smoothness
Skin fine lines | 9 weeks
  Dermatologist grading of skin fine lines
Skin softness | 9 weeks
  Dermatologist grading of skin softness
Skin hydration | 9 weeks
  Dermatologist grading of skin hydration
Skin translucency | 9 weeks
  Dermatologist grading of skin translucency
Pimple | 9 weeks
  Dermatologist grading of pimple
Clogged pores | 9 weeks
  Dermatologist grading of clogged Pores

CONTACTS AND LOCATIONS:
Overall Officials: Chao Yuan, Principal Investigator — Shanghai Skin Disease Hospital
Locations (1):
- Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=12414&filename=Report%20synopsis%20of%20HB%208-week%20HUT.pdf